CLINICAL TRIAL: NCT06655168
Title: Orotracheal Intubation in Newborns: Videolaryngoscopy Vs Direct Laryngoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Mehdi Trifa, Head of Anesthesia and Intensive Care Department, Tunis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 212023
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: The Time Taken for Successful Tracheal Intubation in Each Technique
Keywords: endotracheal intubation, newborn, direct laryngoscopy,video laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video laryngoscopy (Other)
  Interventions: Device: Video Laryngoscopy
- Direct laryngoscopy (Other)
  Interventions: Device: Direct Laryngoscopy

INTERVENTIONS:
Device: Video Laryngoscopy — orotracheal intubation by C-Mac ( Video laryngoscopy)
  Arms: Video laryngoscopy
Device: Direct Laryngoscopy — Orotracheal intubation using Direct Laryngoscopy
  Arms: Direct laryngoscopy

SUMMARY:
The children were randomized into two groups to receive orotracheal intubation after anesthetic induction with neuromuscular blockade, either by direct laryngoscopy (DL, DL group) or by C-MAC video laryngoscopy (VL group)

DETAILED DESCRIPTION:
prospective randomized study including newborns , requiring orotracheal intubation for surgery or mechanical ventilation in the intensive care unit. The children were randomized into two groups to receive orotracheal intubation after anesthetic induction with neuromuscular blockade, either by direct laryngoscopy (DL, DL group) or by C-MAC video laryngoscopy (VL group).

ELIGIBILITY:
Inclusion Criteria:

* newborns requiring orotracheal intubation for surgery or mechanical ventilation in the intensive care unit

Exclusion Criteria:

* age> 01 month

Ages: 1 Minute to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Estimated)
Dates: Start 2023-12-17 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
time taken for successful tracheal intubation | during intubation

SECONDARY OUTCOMES:
the need for additional device | during intubation
the number of attempts | during intubation
Complications during intubation | during intubation
  complications such as desaturation and selective intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Bechir Hamza hospital, Tunis, Tunis Governorate, Tunisia